CLINICAL TRIAL: NCT07371741
Title: PICS Clinic Attendance and Recovery Engagement (PICS-CARE)
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - University Berlin, Charite University, Berlin, Germany
Other Study IDs: PICS-CARE
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Post-intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care unit patients: Intensive care unit patients, which are invited in the post-intensive care outpatient clinic

SUMMARY:
To identify relevant factors influencing attendance at appointments at the PICS outpatient clinic after intensive care treatment in order to derive targeted measures to increase the participation rate or send more targeted invitations.

DETAILED DESCRIPTION:
This retrospective study examines which factors influence patient attendance at structured follow-up appointments after intensive care treatment in the PICS outpatient clinic at Charité. The focus is on analyzing demographic, clinical, and care-related factors that influence actual participation in follow-up care after intensive care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, between January 1, 2021, and December 31, 2025:
* were invited for follow-up care by the PICS outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK)
* were ≥18 years old at the time of the appointment.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care unit patients, who were invited for follow-up care by the PICS outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Follow-up appointment | 01.01.2021- 31.12.2025
  Participation in the first scheduled follow-up appointment at the post-intensive care syndrome (PICS) outpatient clinic (binary: attended vs. did not attend) is measured by medical record review.

SECONDARY OUTCOMES:
Cancellation of a scheduled follow-up appointment. | 01.01.2021- 31.12.2025
  Cancellation of a scheduled follow-up appointment is measured by medical record review.
Reasons for canceling a scheduled appointment. | 01.01.2021- 31.12.2025
  Reasons for canceling a scheduled appointment is measured by medical record review.
Failure to attend a scheduled follow-up appointment. | 01.01.2021- 31.12.2025
  Failure to attend a scheduled follow-up appointment is measured by medical record review.
Death after discharge from the intensive care unit until the first follow-up appointment. | 01.01.2021- 31.12.2025
  Death after discharge from the intensive care unit until the first follow-up appointment is measured by medical record review.
Death between the first and second follow-up appointments. | 01.01.2021- 31.12.2025
  Death between the first and second follow-up appointments is measured by medical record review.
Scheduling a second follow-up appointment after initial presentation at the outpatient clinic. | 01.01.2021- 31.12.2025
  Scheduling a second follow-up appointment after initial presentation at the outpatient clinic is measured by medical record review.
Attendance at the second scheduled follow-up appointment after initial presentation at the outpatient clinic. | 01.01.2021- 31.12.2025
  Attendance at the second scheduled follow-up appointment after initial presentation at the outpatient clinic is measured by medical record review.
Scheduling a third follow-up appointment after initial presentation at the outpatient clinic. | 01.01.2021- 31.12.2025
  Scheduling a third follow-up appointment after initial presentation at the outpatient clinic is is measured by medical record review.
Attendance at the third scheduled follow-up appointment after initial presentation at the outpatient clinic. | 01.01.2021- 31.12.2025
  Attendance at the third scheduled follow-up appointment after initial presentation at the outpatient clinic is measured by medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No